CLINICAL TRIAL: NCT02990598
Title: Hydoxyurea Exposure in Lactation: A Pharmacokinetics Study (HELPS)
Brief Title: Hydoxyurea Exposure in Lactation A Pharmacokinetics Study (HELPS)
Acronym: HELPS
Status: Completed | Type: Observational
Sponsor: Children's Hospital Medical Center, Cincinnati (Other)
Responsible Party: Sponsor
Other Study IDs: 2016-7590_HELPS
Record Dates: First submitted 2016-12-09; First posted 2016-12-13 (Estimated); Last update posted 2019-08-26 (Actual); Status verified 2019-08

CONDITIONS: Sickle Cell Anemia
Keywords: Hydroxyurea
MeSH Terms: conditions — Anemia, Sickle Cell

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — 1. To obtain blood, urine, and breastmilk samples for pharmacokinetics calculations using a scheduled collection and analysis strategy. 2. To calculate distribution ratios for hydroxyurea across compartments, especially plasma to milk; and 3. To create population PK profiles for hydroxyurea to help calculate potential infant drug exposure
Oversight: Data Monitoring Committee: No

SUMMARY:
To examine the pharmacokinetics and distribution of oral hydroxyurea when administered as a single dose to lactating women

ELIGIBILITY:
Inclusion Criteria:

* Lactating females, ≥ 18.0 years of age, at the time of enrollment
* Willingness to limit the baby's exposure to hydroxyurea through breastmilk, such as healthy volunteers using the "pump and dump" technique or avoiding direct breastfeeding or collection of pumped milk for at least 8 hours after taking the hydroxyurea dose. This applies only to healthy controls or women with sickle cell who are not already taking hydroxyurea. Women with sickle cell already taking hydroxyurea may continue to breastfeed their infants.

Exclusion Criteria:

* Persons with known allergies to hydroxyurea
* Failure to sign informed consent, or inability to undergo informed consent process
* Persons for whom it is not feasible or medically advisable to obtain the specimens necessary for this study

Ages: 18 Years to 99 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Healthy Controls and Women taking Hydroxyurea prescribed by treating physician and lactating
Sampling Method: Non-Probability Sample
Enrollment: 16 (Actual)
Dates: Start 2017-03-20 (Actual); Primary Completion 2018-06-19 (Actual); Study Completion 2018-06-19 (Actual)

PRIMARY OUTCOMES:
Hydroxyurea Concentration | 31-Dec-2019
  Hydroxyurea concentration for each collected specimen will be analyzed and summarized.

CONTACTS AND LOCATIONS:
Overall Officials: Russell Ware, MD, PhD, Principal Investigator — Children's Hospital Medical Center, Cincinnati
Locations (1):
- Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio, United States

IPD SHARING:
Plan to Share IPD: No